CLINICAL TRIAL: NCT05420337
Title: Analgesic Effect of Morphine Added to Transverses Abdominis Plane Block; Is it Systemic or Regional Effect?
Brief Title: Analgesic Effect of Morphine Added to Transverses Abdominis Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Meryem Onay, Specialist Doctor-Anesthesiologist, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ESOGU 3
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Pain, Postoperative; Postoperative Complications
Keywords: postoperative pain; transversus abdominis plane block; morphine
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Group I: TAP block with bupivacain and morphine intramuscular will be applied at the end of the operation. Patients will receive paracetamol 1gr 30 minutes before the end of the operation. All patients will undergo IV morphine patient-controlled analgesia (PCA). Pain, opioid consumption, hemodynamic parameters and complications will be monitored in the first 24 hours in the postoperative period.
  Group T: TAP block with bupivacain and morphine will be applied at the end of the operation. Patients will receive paracetamol 1gr 30 minutes before the end of the operation. All patients will undergo IV morphine patient-controlled analgesia (PCA). Pain, opioid consumption, hemodynamic parameters and complications will be monitored in the first 24 hours in the postoperative period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In the postoperative period, the effectiveness and safety of the block will be evaluated by another researcher (blind) who does not know which group the patient is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Intramuscular (Active Comparator): Transversus Abdominis Plane Block will administer with 20 ml of % 0.25 bupivacaine and 0.1 mg/kg morphine intramuscular
  Interventions: Procedure: Group ıntramuscular
- Group TAP (Active Comparator): Transversus Abdominis Plane Block will administer with 20 ml of % 0.25 bupivacaine and 0.1 mg/kg morphine
  Interventions: Procedure: Group TAP

INTERVENTIONS:
Procedure: Group ıntramuscular — Group I will be applied 20 ml of % 0.25 bupivacain internal oblique and transversus abdominis muscle and 0.1 mg/kg morphine ıntramuscular. The blocks will be administered under general anesthesia in supine position by the same anesthesiologist.
  Other Names: Fascial plane block and ıntramuscular morphine at lower abdominal surgery
  Arms: Group Intramuscular
Procedure: Group TAP — Group T will be applied 20 ml of % 0.25 bupivacain and 0.1 mg/kg morphine internal oblique and transversus abdominis muscle. The blocks will be administered under general anesthesia in supine position by the same anesthesiologist.
  Other Names: Fascial plane block with morphine at lower abdominal surgery
  Arms: Group TAP

SUMMARY:
Postoperative pain is a condition that increases morbidity and mortality. Therefore, multimodal analgesia techniques with fascial plan blocks are frequently used.TAP block provides analgesia in the anterior abdominal wall by applying local anesthetic to the fascia between the internal oblique and transversus abdominis muscle. Opioids can be added to local anesthetics to increase the quality and duration of analgesia. The investigators aim is comparasion of TAP block with bupivacaine added morphine and TAP block with bupivacaine plus intramuscular morphine effects on postoperative pain score, total opioid consumption and systemic effects in lower abdominal surgery

DETAILED DESCRIPTION:
At the end of the operation, patients will be randomly divided into 2 groups as Group I (Intramuskuler) and Group T (TAP block). The blocks will be administered under general anesthesia in supine position by same anesthesiologist. Group I (Intramuskuler) will be applied 20 ml of %0.25 bupivacaine between the internal oblique and transversus abdominis muscle and 0.1 mg/kg (ideal body weight) morphine to be performed intramuscular. Group T will be applied 20 ml of %0.25 bupivacaine and 0.1 mg/kg morphine (ideal body weight) between the internal oblique and transversus abdominis muscle. At the end of the operation, the patients with a Modified aldreate score ≥9 will be sent from the postoperative anesthesia unit. All patients will be equipped with an IV morphine patient-controlled analgesia (PCA) device. The solution will be prepared such that morphine is 0.5 mg / ml. PCA 1mg bolus dose will be delivered with 10 min lock-out time. In the postoperative period, the patient was evaluated by another researcher who blind to the groups at the 1st and 6th, 12th and 24th hours. Visual pain scores (VAS) in rest and movement, hemodynamic values, morphine consumption, nausea-vomiting score, itching, ramsey sedation scale, length of hospital stay and postoperative complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Lower abdominal gynecological surgery

Exclusion Criteria:

* Patients with a known allergy to the study drugs,
* Significant cardiac, respiratory, renal or hepatic diseases,
* Bleeding diathesis
* Those with psychiatric illnesses that would interfere with perception and assessment of pain were excluded from this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Comparasion of TAP block with bupivacaine added morphine and TAP block with bupivacaine plus intramuscular morphine effects on postoperative pain score and total opioid consumption in lower abdominal surgery | 24 hours
  Visual analog scale at rest and movement (0 (no pain)-10 (unbearable pain)) Total morphine patient control analgesia prepared 0.5 mg / ml. PCA 1mg bolus dose will be delivered with 10 min lock-out time. Follow up morphine consumption at postoperative 24 hours.

SECONDARY OUTCOMES:
Systemic effects | 24 hours
  Hemodynamic changes, nausea-vomiting (1-none, 2-mild, 3-moderate, 4-severe), itching (1-none, 2-mild, 3-moderate, 4-severe) and ramsay sedation scale systemic effects will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Onay, Principal Investigator — Eskisehir Osmangazi University Faculty Of Medicine
Locations (1):
- Eskisehir Osmangazi University Hospital, Eskişehir, Turkey (Türkiye)

REFERENCES:
- [Background] El Sherif FA, Mohamed SA, Kamal SM. The effect of morphine added to bupivacaine in ultrasound guided transversus abdominis plane (TAP) block for postoperative analgesia following lower abdominal cancer surgery, a randomized controlled study. J Clin Anesth. 2017 Jun;39:4-9. doi: 10.1016/j.jclinane.2017.03.009. Epub 2017 Mar 10. PMID 28494906
- [Background] Chen Q, Liu X, Zhong X, Yang B. Addition of dexmedetomidine or fentanyl to ropivacaine for transversus abdominis plane block: evaluation of effect on postoperative pain and quality of recovery in gynecological surgery. J Pain Res. 2018 Nov 16;11:2897-2903. doi: 10.2147/JPR.S178516. eCollection 2018. PMID 30532583
- [Background] Tsai HC, Yoshida T, Chuang TY, Yang SF, Chang CC, Yao HY, Tai YT, Lin JA, Chen KY. Transversus Abdominis Plane Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:8284363. doi: 10.1155/2017/8284363. Epub 2017 Oct 31. PMID 29226150
- [Background] Abdallah FW, Laffey JG, Halpern SH, Brull R. Duration of analgesic effectiveness after the posterior and lateral transversus abdominis plane block techniques for transverse lower abdominal incisions: a meta-analysis. Br J Anaesth. 2013 Nov;111(5):721-35. doi: 10.1093/bja/aet214. Epub 2013 Jun 27. PMID 23811424
- [Background] Sehgal N, Smith HS, Manchikanti L. Peripherally acting opioids and clinical implications for pain control. Pain Physician. 2011 May-Jun;14(3):249-58. PMID 21587328
- [Derived] Onay M, Kaya O, Telli E, Bilir A, Gulec MS. Are the Analgesic Effects of Morphine Added to Transversus Abdominis Plane Block Systemic or Regional? A Randomized Clinical Trial. Pain Res Manag. 2025 Mar 12;2025:9187270. doi: 10.1155/prm/9187270. eCollection 2025. PMID 40109499